CLINICAL TRIAL: NCT01519180
Title: Study of the Antro-pyloro-duodenal Motor Dysfunction in Idiopathic Gastroparesis
Brief Title: Antro-pyloro-duodenal Motility in Idiopathic Gastroparesis
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2010/148/HP
Record Dates: First submitted 2012-01-18; First posted 2012-01-26 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Gastroparesis
Keywords: gastroparesis; gastric emptying; antro-duodenal manometry
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control group: Healthy volunteers
- Idiopathic gastroparesis: Idiopathic gastroparesis

SUMMARY:
Impaired gastric emptying may cause dyspeptic symptoms including nausea, vomiting and even nutritionnal impairment. Delay in gastric emptying may result from antro-pyloro-duodenal motility impairement.

DETAILED DESCRIPTION:
The aim of this study is therefore to measure antro-pyloro-duodenal motor activity in patients with idiopathic gastroparesis.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic gastroparesis or healthy volunteers
* Idiopathic gastroparesis must have delayed gastric emptying shown using C13 breath test

Exclusion Criteria:

* Diabetic or post-surgical gastroparesis
* Treatment modifying GI motility (prokinetics, opioids...)
* Parkinson or neurologic disease
* Evoluting inflammatory process or neoplasia
* Treatment modifying coagulation
* Patients not affiliated to the French healthcare insurance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Idiopathic gastroparesis and healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2012-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
antro-pyloro-duodenal pressure | 3h
  the main outcome is the pressure measured using pressure sensors within the antrum, the pylorus, and the first part of the duodenum. This will be measured during 3h fast. Pressures measured in the antrum, the pylorus, and the duodenum wiil be compared between healthy volunteers and gastroparetic patients

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Gourcerol, MD, PhD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Service de Physiologie, Rouen, Haute Normandie, France

REFERENCES:
- [Derived] Soliman H, Wuestenberghs F, Desprez C, Leroi AM, Melchior C, Gourcerol G. Physiological characterization of gastric emptying using high-resolution antropyloroduodenal manometry. Am J Physiol Gastrointest Liver Physiol. 2024 Jan 1;326(1):G16-G24. doi: 10.1152/ajpgi.00101.2023. Epub 2023 Oct 24. PMID 37874655